CLINICAL TRIAL: NCT04007081
Title: Salivary Gland Autotransplantation of Marrow Mesenchymal Stromal Cells for Treatment of Radiation-induced Xerostomia - FDA IND (Investigational New Drug) Enabling Studies
Brief Title: Salivary Gland Autotransplantation for Treatment of XRT Induced Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UW19009; 2019-0497 (Other: Institutional Review Board); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); A533300 (Other: UW Madison); Protocol Version 7/24/2020 (Other: UW Madison)
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Xerostomia; Head and Neck Cancer
Keywords: Dry Mouth; MSC; mesenchymal stem cells; adult stem cells; head and neck cancer; salivary gland; radiation; HNC
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Xerostomia (Experimental): Salivary sample collection, quality of life survey, salivary gland imaging, bone marrow aspiration
  Interventions: Procedure: Bone Marrow Aspiration; Diagnostic Test: Ultrasound Imaging of Salivary Glands; Other: Salivary Assay; Other: Quality of Life Instruments

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — collection of approximately 40 mL of bone marrow aspirate
  Other Names: Bone Marrow Collection
Diagnostic Test: Ultrasound Imaging of Salivary Glands — Salivary gland size will be measured by ultrasound.
Other: Salivary Assay — Whole saliva production rates (sialometry) will be measured under unstimulated (first passive drool method) and stimulated (chewing gum) saliva collection conditions
  Other Names: sialometry
Other: Quality of Life Instruments — Participants will self-assess with the following Quality of Life (QoL) surveys: University of Michigan Xerostomia related quality of life scale (XeQOL), the MD Anderson Dysphagia Index (MDADI), and the VAS xerostomia questionnaire.

SUMMARY:
Xerostomia, or dry mouth, is a common side effect of head neck radiation. Current treatment options for radiation-induced xerostomia are generally supportive in nature. Most of these supportive interventions do not reverse xerostomia and are palliative in intent.

The investigators propose that autotransplantation of marrow-derived mesenchymal stromal cells (MSCs) in salivary glands post-RT or post-chemoradiation therapy (CRT) may provide an innovative remedy to treat xerostomia and restore quality of life.

Participants can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
This feasibility study will analyze the salivary composition, salivary viscoelasticity, salivary gland US, and QoL surveys of participants without head and neck cancer (HNC) to determine standard values. The investigators will then compare this to the salivary composition and viscoelasticity of participants with treated HNC.

Additionally, the investigators will examine the paracrine factors of marrow MSCs in order to prove a hypothesis that paracine factors constitutively expressed by marrow MSCs [Wnts, fibroblast growth factors (FGFs), GDNF and others] will directly influence the biology of dormant salivary gland stem cells following intraglandular transplantation and allow for functional recovery following RT.

Primary Objective

* To determine the feasibility of in vitro expansion of marrow-derived MSCs from HNC patients to >50 million cells.

Secondary Objectives

* To assess the stability of salivary function in HNC patients using quality-of-life (QoL) questionnaires and salivary composition analysis.
* To assess the stability of salivary gland size as measured by ultrasound.

Correlative Objectives

* To compare assess the secretome profile of MSCs from HNC patients treated with radiation or, chemoradiation, or previously untreated.
* To compare the salivary composition, viscoelasticity, salivary gland ultrasound, and QoL of HNC patients to non-HNC patients

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥2 years from completion of chemoradiation therapy or radiation therapy (N=6) with subjective complaint of xerostomia or with no diagnosis of HNC (N=5)
* Karnofsky ≥ 60, participant eligible for bone marrow aspirate with wakeful anesthesia
* Not pregnant
* Willing and able to give informed consent
* non-HNC participants only need to meet the following applicable inclusion criteria

  * No history of radiation to the salivary glands
  * Willing and able to give informed consent

Exclusion Criteria:

* Salivary gland disease (e.g., sialolithiasis)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Number of Participant's whose Marrow-Derived MSCs Can be Expanded in vitro to > 50 million cells within two weeks | Up to 1 day to collect, subsequently cultured in vitro for up to 2 weeks
  The feasibility of in vitro expansion of MSCs derived from marrow aspirates collected from participants will be determined by if they can be culture expanded for up to two weeks to generate >50 million MSCs per donor. Feasibility will reported as the number of participants whose marrow-derived MSCs can be expanded in vitro to > 50 million cells within two weeks.

SECONDARY OUTCOMES:
Change in participant QoL: XeQOL | baseline and up to 6 months
  The University of Michigan Xerostomia related quality of life scale (XeQOL) is a 15-item questionnaire about how a participants oral health affects their life. Each item is scored from 1-5 either 'not at all', 'a little', 'somewhat', 'quite a bit', or 'very much' for a total score of 15-75. Higher scores represent greater degree of symptoms.
Change in participant QoL: MDADI | baseline and up to 6 months
  The MD Anderson Dysphagia Inventory (MDADI) is a 20-item questionnaire about how a participants perceive their swallowing ability. Each item is scored from 'strongly agree', 'agree', 'no opinion', 'disagree', or 'strongly disagree'. One question provides a 'global score between 1-5 where 1 is extremely low functioning and 5 is high functioning. The remaining 19 questions measure a composite score from 20-100 where higher scores represent higher degree of function.
Change in participant QoL: VAS | baseline and up to 6 months
  The Visual Analogue Scale (VAS) - xerostomia questionnaire is an 8-item questionnaire about how a participant perceives their dry mouth. Each item is visually scored on a sliding scale (100mm in length) between two extremes (Q1 and Q2 from 'not difficult at all' to 'very difficult', Q3 from 'A lot' to 'None', Q4-Q7 from 'Not Dry at All' to 'Very Dry', and Q8 from 'Not Thirsty at All' to 'Very Thirsty'. The participant places a line on the scale to mark their answer. Change between various time points can be determined based on measured distance along the scale for each answer.
Change in participant Salivary Function: Unstimulated | baseline and up to 6 months
  Unstimulated saliva production will be measured at two time points by the passive drool method over a 5-minute time frame. Participants will allow saliva to pool in the mouth and, then, with head tilted forward, gently guide saliva into a saliva collection aid attached to a cryovial. Difference in weight of the cryovial empty and after the test will represent the amount of saliva produced.
Change in participant Salivary Function: Stimulated | baseline and up to 6 months
  Stimulated saliva production will be measured at two time points by having participants chew inert gum base to the pace of a metronome (70 beats per minute) while expectorating saliva (without swallowing) into the saliva collection aid for 5 minutes total. Difference in weight of the cryovial empty and after the test will represent the amount of saliva produced.
Change in participant Salivary Gland Size | baseline and up to 6 months
  The size of salivary glands will be measured via ultrasound at baseline and up to 6 months on study.

OTHER OUTCOMES:
Compare Secretome Profile of MSCs Between Participant Groups: ELISA | up to 6 months
  The secretome profile of MSCs from HNC participants treated with radiation, chemoradiation, or previously untreated will be statistically compared using enzyme-linked immunosorbent assay (ELISA).
Compare Secretome Profile of MSCs Between Participant Groups: Western Blot | up to 6 months
  The secretome profile of MSCs from HNC participants treated with radiation, chemoradiation, or previously untreated will be statistically compared using and western blots.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Kimple, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/